CLINICAL TRIAL: NCT00150020
Title: Safety and Tolerability of Enteric-Coated Mycophenolate Sodium in Renal Transplant Patients With GI Intolerance
Brief Title: Safety and Tolerability of Enteric-Coated Mycophenolate Sodium (EC-MPS) in Renal Transplant Patients With GI Intolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: novartis, novartis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AUS02
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Renal Transplantation
Keywords: Renal/Kidney; Transplantation; MPA; EC-MPS; Renal Transplantation Patients with GI Intolerance with MMF

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (EC-MPS)

SUMMARY:
The aim of this study is to evaluate the safety and tolerability of EC-MPS in maintenance renal transplant patients who experience gastrointestinal (GI) intolerance due to adverse events associated with mycophenolate mofetil (MMF) and were converted to EC-MPS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-75 years.
2. Recipients of first or secondary cadaveric, living unrelated or living related kidney transplant.
3. Recipients who are at least 4 weeks post renal transplantation.
4. Patients currently receiving MMF (all dosages are allowed), cyclosporine microemulsion, its generic equivalent, cyclosporine USP (modified) or tacrolimus with or without corticosteroids as part of their immunosuppressive regimen for at least 2 weeks.
5. Patients with mild and/or moderate GI complaints (e.g. upper abdominal pain, dyspepsia, anorexia, nausea, vomiting) with or without diarrhea.

Exclusion Criteria:

1. Multi-organ patients (e.g. kidney and pancreas) or previous transplant with any other organ different from kidney (secondary kidney transplant is allowed).
2. Evidence of graft rejection, treatment of acute rejection or unstable renal function within 4 weeks prior to baseline visit.
3. Patients who have received an investigational immunosuppressive drug within 4 weeks prior to study entry.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Tolerability of EC-MPS in combination with CsA-ME or tacrolimus as determined by gastrointestinal symptom rating scale (GSRS) after conversion from MMF in maintenance renal transplant patients with GI intolerance | within 3 months

SECONDARY OUTCOMES:
Safety of EC-MPS in combination with CsA-ME or tacrolimus as determined by incidence and severity of GI adverse events | within 3 months
Tolerability of EC-MPS in combination with CsA-ME or tacrolimus as determined by gastrointestinal symptom rating scale (GSRS) | within 1 month
Efficacy of EC-MPS in combination with CsA-ME or tacrolimus as measured by the incidence of biopsy-proven acute rejection | within 3 months
Tolerability of EC-MPS in combination with CsA-ME or tacrolimus by comparing the two study groups | after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Bolin P, Tanriover B, Zibari GB, Lynn ML, Pirsch JD, Chan L, Cooper M, Langone AJ, Tomlanovich SJ. Improvement in 3-month patient-reported gastrointestinal symptoms after conversion from mycophenolate mofetil to enteric-coated mycophenolate sodium in renal transplant patients. Transplantation. 2007 Dec 15;84(11):1443-51. doi: 10.1097/01.tp.0000290678.06523.95. PMID 18091520